CLINICAL TRIAL: NCT00569062
Title: A Randomized, Double Blind, Placebo Controlled Study to Explore the Antidepressant Properties of P38a Kinase Inhibitor GW856553X 15mg Compared to PBO in Subjects With Major Depressive Disorder Exhibiting Symptoms of Loss of Energy and Interest and Psychomotor Retardation, for a Six Week Treatment Period
Brief Title: A Study of GW856553X For the Treatment of Depression
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Negative data from a GSK PoC study in RA combined with evidence of greater sensitivity of toll-like receptor pathways to p38 inhibition.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PKI108574
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Depressive Disorder, Major
Keywords: Psychomotor retardation; cytokines; GW856553; Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major; Psychomotor Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): GW856553X 7.5mg BID for 6 weeks
  Interventions: Drug: GW856553X
- Placebo (Placebo Comparator): Placebo to match, BID, 6 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GW856553X — GW856553X 7.5mg BID for 6 weeks
  Arms: Arm 1
Other: Placebo — Placebo to match GW856553X
  Arms: Placebo

SUMMARY:
GW856553 is a novel compound, currently in development for the treatment of Major Depressive Disorder (MDD), and other indications. GW856553 inhibits a protein which is responsible for the production of some pro-inflammatory molecules, called cytokines. Increased blood levels of these molecules were seen in populations of MDD patients and this was more apparent in subjects with severe symptoms, psychomotor retardation and loss of energy. Aim of the present study is to assess whether GW856553, by inactivating this protein, is able to suppress the production of the cytokines, and ultimately relieving depression symptoms. In this study GW856553 or placebo is given to MDD patients 7.5md twice daily for 6 weeks.

DETAILED DESCRIPTION:
A randomised, double-blind, placebo-controlled study to explore the antidepressant properties of the P38a kinase inhibitor GW856553X 15mg compared to placebo in subjects with Major Depressive Disorder exhibiting symptoms of loss of energy and interest, and psychomotor retardation, for a six week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female = 18 years of age and < 60 years,
* routine laboratory results within normal ranges,
* Body Mass Index within the range 18.5-35.0 kg/m2 inclusive.
* Subject must have had at least one previous major depressive episode with a diagnosis of MDD in his/her history, and had a successful pharmacological treatment of that episode, and is currently experiencing a recurrence of MDD presently un-medicated.
* Subjects must met the diagnosis of an episode of Major Depressive Disorder in the past 12 weeks but not greater than 24 months.

Exclusion Criteria:

* The subject has any history of liver disease.
* The subject has significant cardiac, pulmonary, metabolic, renal, hepatic or gastrointestinal conditions that, in the opinion of the investigator and/or GSK medical monitor, places the subject at an unacceptable risk as a participant in this trial.
* The subject has a history of autoimmune diseases.
* The subject has any active infectious diseases, including active tuberculosis or a history of active tuberculosis.
* The subject has a history of malignancy, except for surgically cured basal cell carcinoma or females with cured cervical carcinoma (> 2 yrs prior).
* The subject has a history of HIV or other immunosuppressive disease.
* The subject has uncontrolled diabetes.
* The subject is pregnant or nursing.
* Subject has no contact with an adult on a daily basis (i.e., subjects who are not living with at least one other adult or subjects who do not have an adult who contacts them on a daily basis).
* Subject has initiated psychotherapy within three months prior to the Screening visit, or plans to initiate psychotherapy during the trial.
* Subject has received electroconvulsive therapy or transcranial magnetic stimulation or vagal nerve stimulation within the six months prior to the Screening.
* The subject is currently receiving a chronic biological or pharmacologic anti-inflammatory therapy; interferon therapy at any dose or did receive them within 6 months prior randomisation.
* Subjects who have donated a unit of blood within the previous month or intends to donate in the month after completing the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-09-12 (Actual); Primary Completion 2008-06-25 (Actual); Study Completion 2008-06-25 (Actual)

PRIMARY OUTCOMES:
Change from Randomization at Week 6 in Bech subscale (6-item of 17-item Hamilton depression rating [HAMD-17] scale) score | Day 1 (Randomization, Week 0) and Week 6
  HAMD is an instrument for evaluating severity of symptoms of depression, was completed by the participant. The instrument used in this study was the 17-item version (HAM-D17). The Bech subscale of the HAMD-17 is composed of 6 identified items out of the 17 items rated in HAMD-17 scale. Each item is rated on either a 3-point scale (0 to 2) or a 5-point scale (0 to 4). The following symptoms were rated on a 5-point scale (0-4): depressed mood, low self-esteem (guilt), work and interests, psychomotor retardation, and anxiety (psychic). The following symptom was rated on a 3-point scale (0-2): somatic symptoms (general). Total score ranged from 0 to 22, with 0 indicating absence of symptoms and a higher score indicating greater severity of symptoms. Randomization value was defined as the assessment done on Day 1 (Week 0). Change from Randomization was calculated by subtracting the Randomization value from the post-Randomization (Week 6) value.
Change from Randomization (Week 0) at Week 6 in Inventory for Depressive Symptomatology-Clinician rated (IDS-C) scale total score | Day 1 (Randomization, Week 0) and Week 6
  The IDS-C is a standardized 30-item, clinician rated scale to assess the severity of a participant's depressive symptoms. The items were rated on a 4-point scale of 0-3, where 0 indicated absence of symptom and higher score indicated greater severity of symptom. In order to calculate the total score of IDS-C, the following procedures were used: either item 11 or 12 were scored; either item 13 or 14 were scored; if both items 11 and 12 (or 13 and 14) were scored, the highest of the items was scored. The total score was obtained by adding the scores of 28 items of the 30 items. Total scores range from 0-84, with a score of 0 indicating no depression and a score of 84 indicating the most severe depression. Randomization value was defined as the assessment done on Day 1 (Week 0). Change from Randomization was calculated by subtracting the Randomization value from the post-Randomization (Week 6) value.
Change from randomization (Week 0) at Week 6 in Quick Inventory of Depressive symptomatology 16 item self report (QIDS-SR16) scale total score | Day 1 (Randomization, Week 0) and Week 6
  The QIDS-SR16 is a 16-item rating scale of depressive symptoms completed by the participant. The items were rated on a 4-point scale of 0-3, where 0 indicated absence of symptom and higher score indicated greater severity of symptom. The total score was obtained by adding the scores of the items of depressed mood, decreased interest, fatigue, guilt, concentration, suicidal ideation, the highest score on any 1 of the 4 sleep items, the highest score on any 1 appetite/weight item and the highest score on either of the 2 psychomotor items. Total scores range from 0-27, with a score of 0 indicating no depression and a score of 27 indicating the most severe depression. Randomization value was defined as the assessment done on Day 1 (Week 0). Change from Randomization was calculated by subtracting the Randomization value from the post-Randomization (Week 6) value.
Change from Randomization (Week 0) at Week 6 in the morning serum levels of the pro-inflammatory biomarkers | Day 1 (Randomization, Week 0) and Week 6
  The pro-inflammatory biomarkers include the cytokines interleukin 6 (IL-6), IL-10, interleukin 2 receptor alpha (IL-2ra) and tumour necrosis factor alpha (TNFα). Increased circulating levels of IL-6 and TNFα were consistently described in populations of participants suffering from MDD during the symptomatic episode. The assessments were done at Week 0, Week 2 and Week 6. Serum samples for the assessment were taken at 8:00-9:00 h (before dosing and safety blood/urine sampling), 10:00-11:00 h and 12:00-13:00 h (+/-30 minutes). Randomization value was defined as the assessment done on Day 1 (Week 0, pre-dose). Change from Randomization was calculated by subtracting the Randomization value from the post-Randomization (Week 6) value.

SECONDARY OUTCOMES:
Number of participants with any Adverse events (AEs), Serious adverse events (SAEs) or Death | Up to Follow-up (Up to 53 days)
  An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition.
Mean Suicidality Tracking Scale (STS) scores over period | Week 0 up to Week 6
  The suicidality assessment throughout the study was made using the STS. The STS is an 8-item checklist, developed from the MINI Tracking, Module C, designed to assess change in suicidality. Individual items are rated on a 5-point scale from 0 (not at all) to 4 (extremely). The total score ranged from 0-32, where 0 indicated absence of symptoms and higher score indicated greater severity of diseases. Each item in the scale started with question of "yes" or "no", where the participants were asked to score themselves if the response was "yes". This assessment was administered by a physician with adequate training in psychiatry. The STS was administered at every Visit.
Number of participants with abnormal chemistry values | Up to Follow-up (Up to 53 days)
  The assessments were done at Week 0, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6 and Follow-up Visit. The following laboratory parameters of clinical chemistry were analyzed: alkaline phosphatase, alanine transaminase (ALT), aspartate transaminase (AST), bilirubin (total, direct and indirect), total protein, blood urea nitrogen (BUN), albumin, glucose, creatinine, gamma-glutamyl transpeptidase (ϒ-GGT), sodium, potassium, chloride, calcium, phosphate, lactate dehydrogenase (LDH), creatine kinase (CK), C-reactive protein (high sensitivity assay), triglycerides, high-density lipoproteins (HDL), low-density lipoproteins (LDL) and total cholesterol. Randomization value was the value at Week 0 (Day 1). Only those parameters for which at least one abnormal value was reported are summarized.
Number of participants with abnormal hematology values | Up to Follow-up (Up to 53 days)
  The assessments were done at Week 0, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6 and Follow-up Visit. The following laboratory parameters of clinical chemistry were analyzed: hemoglobin, hematocrit, red blood cells (RBC), reticulocytes, platelets, total white blood cells (WBC), total neutrophils, lymphocytes, monocytes, eosinophils, basophils, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH) and mean cell hemoglobin concentration (MCHC). Randomization value was the value at Week 0 (Day 1). Only those parameters for which at least one abnormal value was reported are summarized.
Number of participants with abnormal urinalysis results | Up to Follow-up (Up to 53 days)
  The assessments were done at Week 0, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6 and Follow-up Visit. The urinalysis parameters of glucose, protein, blood and ketones by dipstick test, RBC, WBC and microscopy (if urine dipstick test was abnormal) for WBC, RBC, hyaline casts, granular casts and cellular casts were assessed. The categories with results of few, moderate, many, 3+, 1-3, few (1-5) and trace is presented. Randomization value was the value at Week 0 (Day 1).
Number of participants of vital signs outside range of Potential Clinical Importance (PCI) | Up to Follow-up (Up to 53 days)
  Vital signs assessment included heart rate (HR), systolic blood pressure (SBP) and diastolic blood pressure (DBP), done whilst the participant was in a sitting position for 5 minutes before each reading. Criteria for vital sign values meeting PCI included: SBP < 85 and > 160 millimeters of mercury (mmHg) and increase or decrease from Baseline >= 20 and >= 40 mmHg; DBP < 45 and > 100 mmHg; HR < 40 and > 110 beats per minute (bpm). Assessments were done at Week 0 (at pre-dose and at 3-4 h post-dose ), Week 1, Week 2 (at pre-dose and at 3-4 h post-dose), Week 3, Week 4 (at post-dose only ), Week 5, Week 6 (at pre-dose and at 3-4 h post-dose) and Follow-up Visit. Randomization value was the value at Week 0 (Day 1). Only those parameters for which at least one value of PCI was reported are summarized.
Number of participants of abnormal electrocardiogram (ECG) values | Up to Follow-up (Up to 53 days)
  Full 12-lead ECGs was recorded whilst the participant was in supine position, using an ECG machine that automatically calculated the HR and measured PR, QRS, QT, QTc (b) intervals (Bazett's correction was applied to QTc measurements). The measurement of ECGs were taken at Week 0, Week 2 and Week 6 at pre-dose around 8.00 h and at 12.00-13.00 h, at about 3-4 h post-dose. At Week 4, measurement was taken post-dose only. Randomization value was defined as the assessment done on Day 1 (Week 0). Abnormal ECG findings both not clinically significant (NCS) and clinically significant (CS) is categorized. If the QTc(b) rised above 430 millisecond (msecs) for males and 450 msecs for females during the study, it was considered as abnormal. Other abnormal ranges of PCI included : PR interval <110 and >220 msec; QRS interval <75 and >110 msec; absolute QTc interval >450 and <=499 msec.
Change from randomization (Week 0) at Week 1, 2, 3, 4 and 5 in Bech subscale (6-item of HAMD-17 scale) score | Day 1 (Randomization, Week 0) up to Week 5
  The HAMD is an instrument for evaluating severity of symptoms of depression, was completed by the participant. The instrument used in this study was the 17-item version (HAM-D17). The Bech subscale of the HAMD-17 is composed of 6 identified items out of the 17 items rated in HAMD-17 scale. Each item is rated on either a 3-point scale (0 to 2) or a 5-point scale (0 to 4). The following symptoms were rated on a 5-point scale (0-4): depressed mood, low self-esteem (guilt), work and interests, psychomotor retardation, and anxiety (psychic). The following symptom was rated on a 3-point scale (0-2): somatic symptoms (general). Total score ranged from 0 to 22, with 0 indicating absence of symptoms and a higher score indicating greater severity of symptoms. Randomization value was defined as the assessment done on Day 1 (Week 0). Change from randomization was calculated by subtracting the randomization value from the individual post-randomization (Week 1, 2, 3, 4 and 5) values.
Change from Randomization (Week 0) at Week 1, 2, 3, 4 and 5 in IDS-C scale total score | Day 1 (Randomization, Week 0) up to Week 5
  The IDS-C is a standardized 30-item, clinician rated scale to assess the severity of a participant's depressive symptoms. The items were rated on a 4-point scale of 0-3, where 0 indicated absence of symptom and higher score indicated greater severity of symptom. In order to calculate the total score of IDS-C, the following procedures were used: either item 11 or 12 were scored; either item 13 or 14 were scored; if both items 11 and 12 (or 13 and 14) were scored, the highest of the items was scored. The total score was obtained by adding the scores of 28 items of the 30 items. Total scores range from 0-84, with a score of 0 indicating no depression and a score of 84 indicating the most severe depression. Randomization value was defined as the assessment done on Day 1 (Week 0). Change from Randomization was calculated by subtracting the Randomization value from the individual post-Randomization (Week 1, 2, 3, 4 and 5) values.
Change from randomization (Week 0) at Week 2 and 4 in QIDS-SR16 scale total score | Day 1 (Randomization, Week 0) up to Week 4
  The QIDS-SR16 is a 16-item rating scale of depressive symptoms completed by the participant. The items were rated on a 4-point scale of 0-3, where 0 indicated absence of symptom and higher score indicated greater severity of symptom. The total score was obtained by adding the scores of the items of depressed mood, decreased interest, fatigue, guilt, concentration, suicidal ideation, the highest score on any 1 of the 4 sleep items, the highest score on any 1 appetite/weight item and the highest score on either of the 2 psychomotor items. Total scores range from 0-27, with a score of 0 indicating no depression and a score of 27 indicating the most severe depression. Randomization value was defined as the assessment done on Day 1 (Week 0). Change from Randomization was calculated by subtracting the Randomization value from the individual post-Randomization (Week 2 and 4) values.
Change from randomization (Week 0) at Week 1, 2, 3, 4, 5 and 6 in HAMD-17 scale total score | Day 1 (Randomization, Week 0) up to Week 6
  HAMD-17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression (symptoms such as depressed mood, work and activities, sleep, suicide, psychomotor agitation/retardation, appetite, sexual interest, anxiety, and somatic symptoms). The items of the HAMD-17 are rated on a scale of 0 to 2 or 0 to 4, and the total score ranges from 0 to 52, where 0 indicates absence of symptom and higher scores indicates more severe symptoms. Randomization value was defined as the assessment done on Day 1 (Week 0). Change from Randomization was calculated by subtracting the Randomization value from the individual post-Randomization (Week 1, 2, 3, 4, 5 and 6) values.
Percentage of participants with Bech subscale (6-item HAMD-17) score responder and remitter at Week 6 | Week 6
  The HAMD is an instrument for evaluating severity of symptoms of depression, was completed by the participant. The Bech subscale of the HAMD-17 is composed of 6 identified items out of the 17 items rated in HAMD-17 scale. Each item is rated on either a 3-point scale (0 to 2) or a 5-point scale (0 to 4). The following symptoms were rated on a 5-point scale (0-4): depressed mood, low self-esteem (guilt), work and interests, psychomotor retardation, and anxiety (psychic). The following symptom was rated on a 3-point scale (0-2): somatic symptoms (general). Total score ranged from 0 to 22, with 0 indicating absence of symptoms and a higher score indicating greater severity of symptoms. Responders were defined as participants with a reduction in total score of >=50% from randomization at Week 6 or study exit. Remitters were defined as participants whose total score was <=4 at Week 6 or study exit. Randomization value was defined as assessment done at Day 1 (Week 0).
Percentage of participants with IDS-C scale total score responder and remitter at Week 6 | Week 6
  The IDS-C is a standardized 30-item, clinician rated scale to assess the severity of a participant's depressive symptoms. The items were rated on a 4-point scale of 0-3, where 0 indicated absence of symptom and higher score indicated greater severity of symptom. In order to calculate the total score of IDS-C, the following procedures were used: either item 11 or 12 were scored; either item 13 or 14 were scored; if both items 11 and 12 (or 13 and 14) were scored, the highest of the items was scored. The total score was obtained by adding the scores of 28 items of the 30 items. Total scores range from 0-84, with a score of 0 indicating no depression and a score of 84 indicating the most severe depression. Responders were defined as participants with a reduction in total score of >=50% from randomization at Week 6 or study exit. Remitters were defined as participants whose total score was <=15 at Week 6 or study exit. Randomization value was defined as assessment done at Day 1 (Week 0).
Percentage of participants with QIDS-SR16 scale total score responder and remitter at Week 6 | Week 6
  The QIDS-SR16 is a 16-item rating scale of depressive symptoms completed by the participant. The items were rated on a 4-point scale of 0-3, where 0 indicated absence of symptom and higher score indicated greater severity of symptom. The total score was obtained by adding the scores of the items of depressed mood, decreased interest, fatigue, guilt, concentration, suicidal ideation, the highest score on any 1 of the 4 sleep items, the highest score on any 1 appetite/weight item and the highest score on either of the 2 psychomotor items. Total scores range from 0-27, with a score of 0 indicating no depression and a score of 27 indicating the most severe depression. Responders were defined as participants with a reduction in total score of >=50% from randomization at Week 6 or study exit. Remitters were defined as participants whose total score was <=5 at Week 6 or study exit. Randomization value was defined as assessment done at Day 1 (Week 0).
Change from Randomization in Psychomotor Retardation subscale of the IDS-C scale over Week 6 | Day 1 (Randomization, Week 0) up to Week 6
  The IDS-C is a standardized 30-item, clinician rated scale to assess the severity of a participant's depressive symptoms. The Psychomotor Retardation subscale IDS-C is determined by a 5 item subscale of the IDS-C: item 5: mood (sad); item 15: concentration/decision making; item 20: energy/fatigability; item 23: psychomotor slowing; Item30: leaden paralysis/physical energy. The items were rated on a 4-point scale of 0-3, where 0 indicated absence of symptom and higher score indicated greater severity of symptom. The total score was obtained by adding the scores of the 5 items. Total scores range from 0-15, with a score of 0 indicating no depression and higher score indicating more severe depression. Randomization value was defined as the assessment done on Day 1 (Week 0). Change from Randomization was calculated by subtracting the Randomization value from the individual post-Randomization (Week 1, 2, 3, 4, 5 and 6) values.
Change from Randomization in Psychomotor Retardation subscale of the QIDS-SR16 scale over Week 6 | Day 1 (Randomization, Week 0) up to Week 6
  The QIDS-SR16 is a 16-item rating scale of depressive symptoms completed by the participant. The Psychomotor Retardation subscale QIDS-SR16 is determined by a 4 item subscale of the QIDS-SR16: depressed mood, decision making, energy, psychomotor slowing. The items were rated on a 4-point scale of 0-3, where 0 indicated absence of symptom and higher score indicated greater severity of symptom. Total scores range from 0-12, with a score of 0 indicating no depression and higher score indicating more severe depression. Randomization value was defined as the assessment done on Day 1 (Week 0). Change from Randomization was planned to be calculated by subtracting the Randomization value from the individual post-Randomization (Week 1, 2, 3, 4, 5 and 6) values. Data for this outcome measure was not collected and hence no result summary was produced during analysis.
Change from Randomization in Psychomotor Retardation-Psychomotor Slowing item 23 of the IDS-C scale over Week 6 | Day 1 (Randomization, Week 0) up to Week 6
  The IDS-C is a standardized 30-item, clinician rated scale to assess the severity of a participant's depressive symptoms. The Psychomotor Retardation-Psychomotor Slowing item 23 of the IDS-C scale was rated on a 4-point scale of 0-3, where 0 indicated absence of symptom and higher score indicated greater severity of symptom. Randomization value was defined as the assessment done on Day 1 (Week 0). Change from Randomization was calculated by subtracting the Randomization value from the individual post-Randomization (Week 1, 2, 3, 4, 5 and 6) values.
Change from Randomization in Psychomotor Retardation-Psychomotor Slowing item 15 of QIDS-SR16 scale over Week 6 | Day 1 (Randomization, Week 0) up to Week 6
  The QIDS-SR16 is a 16-item rating scale of depressive symptoms completed by the participant. The Psychomotor Slowing item 15 of QIDS-SR16 scale was rated on a 4-point scale of 0-3, where 0 indicated absence of symptom and higher score indicated greater severity of symptom. Randomization value was defined as the assessment done on Day 1 (Week 0). Change from Randomization was calculated by subtracting the Randomization value from the individual post-Randomization (Week 2, 4 and 6) values.
Functional assessment of Fatigue and Sleepiness over Week 6 | Day 1 (Randomization, Week 0) up to Week 6
  The Fatigue question is derived from the Functional Assessment of Chronic Illness Therapy- Fatigue (FACIT-F) questionnaire. The Sleepiness question is derived from the epidemiologic questionnaire used to identify Excessive Daytime Sleepiness (EDS) in a general population and in individual suffering from depression. Questions were planned to be asked by the Investigator or designee for fatigue as "Did you feel fatigued or tired during the past 7 days?"; for sleepiness as "In the past 7 days, did you either feel sleepy during the day (but managed to stay awake) or have an irresistible sleep attack during the day, or both?" The questions are scored on a 5-point scale of 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much. The score ranged from 0-5, where 0 indicated absence of symptom and higher score indicated greater severity of symptom. Data for this outcome measure was not collected and hence no result summary was produced during analysis.
Change from Randomization in Visual Analogue Scale (VAS) of Fatigue/Tiredness and Sleepiness (at time of cytokine sampling) over Week 6 | Day 1 (Randomization, Week 0) up to Week 6
  Four different VAS (0-100 millimeter, minimum-maximum) for Sleepiness and Fatigue/Tiredness was scored before cytokine sampling at pre-dose, 2 h and 4 h post-dose. VAS score for Sleepiness and Fatigue/Tiredness consist of following: item 1: alert (0=alert, 100=drowsy); item 2: sleepy (0=sleepy, 100=awake); item 3: strong (0=strong, 100=feeble); item 4: most tired ever felt (0=most tired ever felt, 100=less tired ever felt). Fatigue/Tiredness was based on score of item 3 and 4 and sleepiness on score of item 1 and 2. All item scores do not move in same direction. Score for item 1 and 3 ranged from 0-100, where 0=absence of symptom and higher score=greater severity of symptom. Score for item 2 and 4 ranged from 0-100, where 0=most severe symptom and higher score=less severe symptom. Randomization value defined as assessment done on Day 1 (Week 0, pre-dose). Change from Randomization was calculated by subtracting Randomization value from individual post-Randomization (Week 0-6) values.
Change from Randomization in Fatigue-Energy item 20 of the IDS-C scale over Week 6 | Day 1 (Randomization, Week 0) up to Week 6
  The IDS-C is a standardized 30-item, clinician rated scale to assess the severity of a participant's depressive symptoms. The Fatigue-Energy item 20 of the IDS-C scale was rated on a 4-point scale of 0-3, where 0 indicated absence of symptom and higher score indicated greater severity of symptom. Randomization value was defined as the assessment done on Day 1 (Week 0). Change from Randomization was calculated by subtracting the Randomization value from the individual post-Randomization (Week 1, 2, 3, 4, 5 and 6) values.
Change from Randomization in Energy/Fatigue item 14 of the QIDS-SR16 scale over Week 6 | Day 1 (Randomization, Week 0) up to Week 6
  The QIDS-SR16 is a 16-item rating scale of depressive symptoms completed by the participant. The Energy/Fatigue item 14 of the QIDS-SR16 scale was rated on a 4-point scale of 0-3, where 0 indicated absence of symptom and higher score indicated greater severity of symptom. Randomization value was defined as the assessment done on Day 1 (Week 0). Change from Randomization was calculated by subtracting the Randomization value from the individual post-Randomization (Week 2, 4 and 6) values.
Change from Randomization in plasma cortisol over Week 6 | Day 1 (Randomization, Week 0) up to Week 6
  The assessments were done at Randomization (Day1, pre-dose, 2 h and 4 h post dose), Week 2 (pre-dose, 2 h and 4 h post-dose) and Week 6 (pre-dose, 2 h and 4 h post-dose). Randomization value was defined as the assessment done on Day 1 (Week 0, pre-dose). Change from Randomization was calculated by subtracting the Randomization value from the individual post-Randomization (Week 0 [2 h and 4 h post dose], Week 2 [pre-dose, 2 h and 4 h post-dose] and Week 6 [pre-dose, 2 h and 4 h post-dose]) values.
Change from Randomization in serum TNFα/IL-10 ratio over Week 6 | Day 1 (Randomization, Week 0) up to Week 6
  The assessments were done at Week 0, Week 2 and Week 6. Serum samples for the assessment were taken at 8:00-9:00 h (before dosing and safety blood/urine sampling), 10:00-11:00 h and 12:00-13:00 h (± 30 minutes). Randomization value was defined as the assessment done on Day 1 (Week 0, pre-dose). Change from Randomization was calculated by subtracting the Randomization value from the individual post-Randomization (Week 0 [2 h and 4 h post-dose], Week 2 [pre-dose, 2 h and 4 h post-dose] and Week 6 [pre-dose, 2 h and 4 h post-dose]) values.
Change from Randomization in high sensitivity C-reactive protein (hs-CRP) over Week 6 | Day 1 (Randomization, Week 0) up to Week 6
  The assessments were done at Week 0, Week 2 and Week 6. Randomization value was defined as the assessment done on Day 1 (Week 0). Change from Randomization was calculated by subtracting the Randomization value from the individual post-Randomization (Week 2 and Week 6) values.
Change from Randomization in number of leukocytes over Week 6 | Day 1 (Randomization, Week 0) up to Week 6
  The assessments were done at Week 0, Week 1, Week 2, Week 3, Week 4, Week 5 and Week 6. Randomization value was defined as the assessment done on Day 1 (Week 0). Change from Randomization was calculated by subtracting the Randomization value from the individual post-Randomization (Week 1 to 6) values.
Plasma concentration of GW856553X and GSK198602 | Pre-dose and 4 h post-dose at Week 2 and Week 6
  Plasma concentration of GW856553X and of the metabolite GSK198602 was assessed during the treatment period. Blood samples were collected at 8:00 h (before dosing) and 12:00-13:00 h (about 4 h after dosing) at Weeks 2 and 6 of the treatment period.
Maximum plasma concentration (Cmax) of GW856553X and GSK198602 | Pre-dose and 4 h post-dose at Week 2 and Week 6
  Plasma concentration of GW856553X and of the metabolite GSK198602 was assessed during the treatment period. Blood samples were collected at 8:00 h (before dosing) and 12:00-13:00 h (about 4 h after dosing) at Weeks 2 and 6 of the treatment period. The first occurrence of the maximum observed plasma concentration was planned to be determined directly from the raw concentration-time data. The data for this outcome measure was not derived due to early termination.
Median time to Cmax (tmax) and the terminal phase half-life (t1/2) | Pre-dose and 4 h post-dose at Week 2 and Week 6
  Plasma concentration of GW856553X and of the metabolite GSK198602 was assessed during the treatment period. Blood samples were collected at 8:00 h (before dosing) and 12:00-13:00 h (about 4 h after dosing) at Weeks 2 and 6 of the treatment period. The time at which Cmax observed was planned to be determined directly from the raw concentration-time data. The apparent t1/2 was planned to be obtained as the ratio of ln2/λz, where λz is the terminal phase rate constant estimated by linear regression analysis of the log transformed concentration-time data. The data for this outcome measure was not derived due to early termination.
The area under the plasma concentration-time curve (AUC) | Pre-dose and 4 h post-dose at Week 2 and Week 6
  Blood samples were collected at 8:00 h (before dosing) and 12:00-13:00 h (about 4 h after dosing) at Weeks 2 and 6 of the treatment period. The AUC was planned to be assessed from time zero (pre-dose) extrapolated to infinite time (AUC0-infinity) and from time zero (pre-dose) to last time of quantifiable concentration within a participant across all treatments (AUC0-t). AUC0-t was planned to be determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations. The AUC0-infinity was planned to be calculated, where data permitted, as the sum of AUC0-t and Ct/z, where Ct is the observed plasma concentration obtained from the log-linear regression analysis of the last quantifiable time-point and z is the terminal phase rate constant. The data for this outcome measure was not derived due to early termination.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- GSK Investigational Site, Tartu, Estonia
- India (5):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Ludhiana
  - GSK Investigational Site, Manipal
  - GSK Investigational Site, Mumbai
  - GSK Investigational Site, Pune
- Russia (4):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Smolensk

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: PKI108574 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: PKI108574 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: PKI108574 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: PKI108574 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: PKI108574 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register